CLINICAL TRIAL: NCT03131193
Title: Estimating the Returns to Provider Human Capital
Brief Title: Primary Care Provider Supply and Patient Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RAND (Other)
Responsible Party: Principal Investigator, Edward Okeke, Policy Researcher, RAND
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: R01HD083444 (NIH)
Record Dates: First submitted 2017-03-10; First posted 2017-04-27 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-10

CONDITIONS: Health Services Accessibility; Health Behavior; Health Care Quality, Access, and Evaluation
MeSH Terms: conditions — Health Behavior | interventions — Physicians

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- No provider - No cash transfer (No Intervention): Study primary health centers (PHC) will carry out business-as-usual, with no additional staffing or changes to usual clinic operations. Study participants who live in the community served by the PHC will not receive any incentives (conditional cash transfer) to encourage them to seek care at the study clinic.
- No Provider - Cash Transfer (Experimental): Study primary health centers (PHC) will carry out business-as-usual, with no additional staffing or changes to usual clinic operations. Study participants who live in the community served by the study PHC will receive a conditional cash transfer if they use services provided by the study PHC.
  Interventions: Behavioral: Conditional Cash Transfer
- Physician - No Cash Transfer (Experimental): Study PHCs will receive an additional health provider - a physician. Study participants who live in the community served by the PHC will not receive any incentives (conditional cash transfer) to encourage them to seek care at the study clinic.
  Interventions: Other: Physician
- Physician - Cash Transfer (Experimental): Study PHCs will receive an additional health provider - a physician. Study participants who live in the community served by the study PHC will receive a conditional cash transfer if they use services provided by the study PHC.
  Interventions: Other: Physician; Behavioral: Conditional Cash Transfer
- Mid-level Provider - No Cash Transfer (Experimental): Study PHCs will receive an additional health provider - a mid-level provider. Study participants who live in the community served by the PHC will not receive any incentives (conditional cash transfer) to encourage them to seek care at the study clinic.
  Interventions: Other: Mid-level provider
- Mid-level Provider - Cash Transfer (Experimental): Study PHCs will receive an additional health provider - a mid-level provider. Study participants who live in the community served by the study PHC will receive a conditional cash transfer if they use services provided by the study PHC.
  Interventions: Other: Mid-level provider; Behavioral: Conditional Cash Transfer

INTERVENTIONS:
Other: Physician — Study primary health centers will be staffed with an additional physician
  Arms: Physician - Cash Transfer; Physician - No Cash Transfer
Other: Mid-level provider — Study primary health centers will be staffed with an additional mid-level provider
  Arms: Mid-level Provider - Cash Transfer; Mid-level Provider - No Cash Transfer
Behavioral: Conditional Cash Transfer — Study participants (who are pregnant women) will receive a cash transfer conditional upon: registering for and attending antenatal care in the study clinic, giving birth in the study clinic and completing a postnatal visit with the new infant
  Arms: Mid-level Provider - Cash Transfer; No Provider - Cash Transfer; Physician - Cash Transfer

SUMMARY:
The evidence on how primary care provider supply and skill relates to patient outcomes is limited and inconclusive. The issue of skill is a particularly important one in low-income countries where the shortage of skilled medical professionals has led to greater use of the task-shifting model in which medical tasks are redistributed from highly skilled health workers to mid-level providers who receive less training. In this large-scale cluster-randomized trial, the investigators randomly select primary health care facilities to receive a highly skilled provider (a doctor), a mid-level health provider, or no additional providers (the control group). The investigators study the effect of this intervention on patient outcomes. Embedded within this trial is another experimental intervention in which pregnant women residing in communities served by the primary health care facilities are assigned to receive a cash transfer conditional on using antenatal, delivery and postnatal care. The investigators study the effect of the cash transfer on health care utilization and on maternal and infant outcomes.

DETAILED DESCRIPTION:
180 primary health care facilities in Nigeria are participating in this study. In one arm of this trial, 60 of the participating facilities are randomly assigned a physician (in addition to existing clinic staff); in a second arm, 60 facilities are randomly assigned an additional mid-level provider (of similar training to existing providers); and the third arm consists of facilities that receive no additional providers (the control group). Assigned providers will practice in those facilities for approximately one year. Stratifying by treatment arm, the investigators further randomize 10-15 enumeration areas within each facility catchment (service) area to either a Conditional Cash Transfer (CCT) arm or to a control arm. The cash transfer is intended for currently pregnant women in those enumeration areas and is conditioned upon attending four antenatal care visits, giving birth in the facility, and attending at least one postnatal visit.

To measure the effects of the interventions the investigators randomly sample 15 households in each facility catchment area and enroll all currently pregnant women within the study enumeration areas. Women at an advanced stage of pregnancy - third trimester - are excluded because such women will not be exposed to the intervention for the majority of their pregnancy. All household members are interviewed at baseline, midline (6 months later) and endline (12 months later) to collect information about health-seeking behavior and health status. Pregnant women are also interviewed at baseline and approximately 1-3 months after birth to collect information about health care utilization and birth outcomes. Additionally the investigators collect data from the participating health facilities and providers. Using a combination of provider surveys, clinical vignettes, direct clinical observation, and patient exit interviews the investigators examine the effects of the intervention on service delivery and quality.

ELIGIBILITY:
Inclusion Criteria for Households:

• Resident in a community served by the study PHC

Exclusion Criteria for Households: none

Inclusion Criteria for Women:

* Resident in a community served by the study PHC
* Must be in 1st or 2nd trimester of pregnancy

Exclusion Criteria for Women:

• 3rd trimester of pregnancy

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 10852 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Clinic attendance | 6-12 months after enrollment
  Utilization of health services will be measured using a questionnaire
Self-reported health | 6-12 months after enrollment
  Self-reported health status will be measured using a questionnaire

SECONDARY OUTCOMES:
Mortality | 6-12 months after enrollment
  Child mortality will be measured using a questionnaire
Quality of care | 6-12 months after enrollment
  Process quality based on adherence to clinical protocols will be measured via direct observation (observer will complete a standardized checklist)
Child weight | 12 months after enrollment
  Child weight in kg will be measured using a weighing scale
Child height | 12 months after enrollment
  Child height in cm will be measured using a measuring board or stadiometer as appropriate

CONTACTS AND LOCATIONS:
Overall Officials: Edward N Okeke, MD, PhD, Principal Investigator — RAND
Locations (1):
- Aminu Kano Teaching Hospital, Kano, Nigeria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Okeke EN, Wagner Z, Abubakar IS. Maternal Cash Transfers Led To Increases In Facility Deliveries And Improved Quality Of Delivery Care In Nigeria. Health Aff (Millwood). 2020 Jun;39(6):1051-1059. doi: 10.1377/hlthaff.2019.00893. PMID 32479220
- [Background] Okeke EN, Abubakar IS. Healthcare at the Beginning of Life and Child Survival: Evidence from a Cash Transfer Experiment in Nigeria. J Dev Econ. 2020 Mar;143:102426. doi: 10.1016/j.jdeveco.2019.102426. Epub 2019 Nov 22. PMID 32863533
- [Background] Okeke EN. Money and my mind: Maternal cash transfers and mental health. Health Econ. 2021 Nov;30(11):2879-2904. doi: 10.1002/hec.4398. Epub 2021 Aug 30. PMID 34462990